CLINICAL TRIAL: NCT01155648
Title: Increasing Pressure Support During Chest Wall Compression is Useful During Respiratory Therapy?
Brief Title: Pressure Support During Chest Wall Compression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Federal University of Rio Grande do Sul, Hospital de Clínicas de Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 07-504
Record Dates: First submitted 2010-06-23; First posted 2010-07-02 (Estimated); Last update posted 2010-07-02 (Estimated); Status verified 2010-06

CONDITIONS: Respiration, Artificial; Critical Care
Keywords: Mechanical ventilation; Chest physiotherapy; Chest wall compression
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PSV group. (Experimental): Chest wall compression plus increase of 10 cmH2O of PSV.
  Interventions: Device: Chest wall compression plus increase of 10 cmH2O in inspiratory pressure during Pressure Support Ventilation for ten minutes in chest.
- chest wall compression group (Active Comparator): Chest wall compression
  Interventions: Device: Chest wall compression for ten minutes in chest

INTERVENTIONS:
Device: Chest wall compression plus increase of 10 cmH2O in inspiratory pressure during Pressure Support Ventilation for ten minutes in chest.
  Arms: PSV group.
Device: Chest wall compression for ten minutes in chest
  Arms: chest wall compression group

SUMMARY:
The purpose of this study is to compare two physiotherapy techniques: chest wall compression versus chest wall compression plus increase of 10 cmH2O in inspiratory pressure.

DETAILED DESCRIPTION:
1. After being placed in the supine position in bed, with head angle elevation at 30°, patients were randomized to:group 1 (G1): chest wall compression for ten minutes in chest or group 2 (G2): chest wall compression plus increase of 10 cmH2O in IP in PSV for ten minutes in chest.
2. Clinical variables and APACHE II were registered.
3. Parameters analyzed at the beginning (1) and at the end (2) of the protocol were: variation of peak pressure (ΔPp=Pp2-Pp1),variation of tidal volume (ΔVT =VT2-VT1), variation of dynamic compliance (ΔCdyn= Cdyn2-Cdyn1).
4. The amount of variation of mucus secretion aspirated (ΔSa= Sa2-Sa1) at the end was also measured

ELIGIBILITY:
Inclusion Criteria:

* Patients on mechanical ventilation over 48 hours
* With ventilatory drive
* Hemodynamically stable MAP> 60 mmHg
* With treatment of respiratory therapy

Exclusion Criteria:

* Contra indication of increased positive inspiratory pressure
* Peak pressure in the upper airway > 40 cmH2O
* Osteoporosis diagnosis
* Deny to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2008-05; Primary Completion 2009-06 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Variation of mucus secretion aspirated. | Two years

SECONDARY OUTCOMES:
Hemodynamic and pulmonary parameters. | Two years
  The hemodynamic and pulmonary parameters were collected: Hart rate (HH), respiratory rate (f), mean arterial pressure (MAP) and peripheral arterial saturation of oxygen (SpO2); peak inspiratory pressure (Ppeak),and Tidal volume (VT) measured in the ventilator, dynamic compliance (Cdyn calculated through the formula VT/ Ppeak - PEEP)

CONTACTS AND LOCATIONS:
Overall Officials: Silvia R Vieira, PhD, Principal Investigator — Federal University of Rio Grande do Sul, Hospital de Clínicas de Porto Alegre
Locations (1):
- Federal University of Rio Grande do Sul, Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] Naue Wda S, Forgiarini Junior LA, Dias AS, Vieira SR. Chest compression with a higher level of pressure support ventilation: effects on secretion removal, hemodynamics, and respiratory mechanics in patients on mechanical ventilation. J Bras Pneumol. 2014 Jan-Feb;40(1):55-60. doi: 10.1590/S1806-37132014000100008. PMID 24626270
- [Derived] Naue Wda S, da Silva AC, Guntzel AM, Condessa RL, de Oliveira RP, Rios Vieira SR. Increasing pressure support does not enhance secretion clearance if applied during manual chest wall vibration in intubated patients: a randomised trial. J Physiother. 2011;57(1):21-6. doi: 10.1016/S1836-9553(11)70003-0. PMID 21402326